CLINICAL TRIAL: NCT03401892
Title: Retinal Neuro-vascular Coupling in Patients With Non-arteritic Anterior Ischemic Optic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Section Head Ophthalmo-Pharmacology, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-210917
Record Dates: First submitted 2018-01-10; First posted 2018-01-17 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Anterior Ischemic Optic Neuropathy
MeSH Terms: conditions — Optic Neuropathy, Ischemic | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with a history of NAION (Experimental): patients with a history of non-arteritic anterior ischemic optic neuropathy (NAION) in one eye
  Interventions: Device: Dynamic Vessel Analyzer (DVA); Device: Fourier Domain Doppler Optical Coherence Tomography (FDOCT); Device: Optical coherence tomography (OCT)
- Healthy control subjects (Experimental): healthy age-and sex- matched control subjects
  Interventions: Device: Dynamic Vessel Analyzer (DVA); Device: Fourier Domain Doppler Optical Coherence Tomography (FDOCT); Device: Optical coherence tomography (OCT)

INTERVENTIONS:
Device: Dynamic Vessel Analyzer (DVA) — Retinal vessel diameters and oxygen saturation will be measured with the DVA device.
Device: Fourier Domain Doppler Optical Coherence Tomography (FDOCT) — Retinal blood flow will be assessed using FDOCT.
Device: Optical coherence tomography (OCT) — Nerve fiber layer thickness and central retinal thickness will be measured using OCT.

SUMMARY:
Ischemic optic neuropathy is among the most common causes of serious impaired vision in the middle-aged and elderly population in the western world. The current study focuses on a subgroup of ischemic optic neuropathy, the so-called non-arteritic ischemic optic neuropathy (NAION). Although the exact pathogenesis of NAION has not been fully clarified it is known that patients with cardio-vascular risk factors such as hypertension, diabetes mellitus and dyslipidemia have also an increased risk to develop NAION. Along this line of thought it has been shown that patients with a history of NAION in one eye have an increased risk to develop NAION also on the contralateral eye. However, clinical studies investigating ocular perfusion abnormalities in patients with NAION are sparse and even contradicting. Thus, the current study seeks to measure ocular blood flow parameters in patients with a history of NAION and compare it to healthy age-matched subjects.

ELIGIBILITY:
Inclusion criteria for healthy subjects:

* Men and women aged over 18 years
* Non-smokers
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropy < 6 Dpt.

Inclusion criteria for patients with NAION:

* Men and women aged over 18 years
* History of NAION in one eye
* Normal ophthalmic findings, ametropy < 6 Dpt.
* Adequate visual acuity to allow participation in the ocular blood flow measurements
* A potential participant has to be on stable doses of all medications he/she is taking because of consisting illnesses according to medical history for at least 30 days prior inclusion, if considered relevant by the investigator.

Any of the following will exclude a healthy subject from the study:

* Current ocular disease or history of NAION
* Presence or history of a severe medical condition as judged by the clinical investigator
* Untreated Arterial hypertension
* History or family history of epilepsy
* Presence of any abnormalities preventing reliable measurements in the study eye as judged by the investigator
* Best corrected visual acuity < 0.5 Snellen
* Ametropy ≥ 6 Dpt
* Pregnancy or planned pregnancy
* Alcoholism or substance abuse

Any of the following will exclude a patient from the study:

* Presence or history of a severe medical condition other NAION as judged by the clinical investigator
* Untreated Arterial hypertension
* History or family history of epilepsy
* Presence of any abnormalities preventing reliable measurements in the study eye as judged by the investigator
* Best corrected visual acuity < 0.5 Snellen in the non-affected eye
* Ametropy ≥ 6 Dpt
* Pregnancy, planned pregnancy
* Alcoholism or substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-06-11 (Actual)

PRIMARY OUTCOMES:
Flicker light induced hyperemia in retinal vessels | 1 day
  Response of retinal vessels to increased neuronal activity assessed with flicker light

SECONDARY OUTCOMES:
Retinal vessel diameters | 1 day
  Response of retinal vessel diameters to flicker light assessed with DVA
Retinal oxygen saturation | 1 day
  Retinal oxygen saturation measured with DVA
Retinal blood flow | 1 day
  Response of retinal blood flow to flicker light assessed with FDOCT
Retinal nerve fiber layer thickness | 1 day
  Retinal nerve fiber layer thickness measured using OCT
Central retinal thickness | 1 day
  Central retinal thickness using OCT

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhöfer, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria